CLINICAL TRIAL: NCT02818933
Title: A Randomized Study of the Automated Self-Administered 24-hour Recall Compared to an Interviewer-administered 24-hour Diet Recall in Adolescents
Brief Title: Diet Intake Estimation of Tweens and Teens: The DIETT Study
Acronym: DIETT
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: CIN_"HughesDIETT"_001
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Diet Intake Assessment
Keywords: 24-hour diet recall; Adolescents; Web-based diet recall

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Aim 1: This group follows a crossover design where adolescents 12-17 years old (n=10) complete a diet recall using one of the two methods (interviewer-administered vs web-based), and then does another diet recall using the other method about a week later. Participants are randomly assigned to the order in which they complete each method of diet recall.
- Aim 2, interviewer-administered recall: This group of adolescents 12-17 years old (n=10) completes an interviewer-administered diet recall once a week for 6 weeks.
- Aim 2, web-based recall: This group of adolescents 12-17 years old (n=10) completes a web-based self-administered diet recall once a week for 6 weeks.

SUMMARY:
The purpose of this pilot study is to assess the quality of self-report data obtained using the Automated Self Administered 24-Hour Recall (ASA24-Kids-2014) relative to an interviewer administered 24-hour recall in a sample of adolescents ages 12-17 years, to determine their method preference, and to assess issues related to each method.

DETAILED DESCRIPTION:
Self-reported dietary intake currently provides the best approach to quantify foods and nutrients for many nutrition research studies. The interviewer administered 24-hour diet recall is generally considered the best available method; however, it is limited by a high degree of participant burden and cost. A web-based, automated, self-administered 24-hour recall (ASA24-Kids-2014) was recently designed by researchers at the National Cancer Institute (NCI) to mimic the interviewer administered 24-hour recall approach to collecting high quality dietary intake data in children and adolescents while minimizing time and cost. Although the ASA24-Kids-2014 is a potentially useful and cost-effective tool for collecting dietary data for research studies in children and adolescents, it has not been validated for use in pediatric populations. A total of 30 adolescents will be recruited to achieve the study aims. For Aim 1, 10 participants will complete one diet recall using ASA24-Kids-2014 and one interviewer administered 24-hour recall. Their feedback on both methods and preference will be assessed. For Aim 2, 20 participants will be randomly assigned to complete six (one per week) web-based or interviewer administered 24-hour recalls. Data from Aim 2 will be analyzed to determine whether the reporting quality decays over time for each method. In addition, feedback from participants in both aims will be collected on specific factors related to the recall methods such as ease of use, technical challenges, flexibility, duration, and database completeness. Results obtained from this pilot study could provide critical information to design a larger method comparison study to rigorously assess the performance of the ASA24-Kids web-based diet recall.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents at least 12 years old and no greater than 17 years old who have access to a phone and a desktop or laptop computer.

Exclusion Criteria:

* Persons having prior experience completing food recalls, either for a research study, or for personal use
* persons having prior experience with mobile food apps, either for research or for personal use
* persons following a special diet
* persons having a mental, physical, or visual limitation that would hinder their ability to use a computer or recall from memory
* Non-English speakers are excluded because using an interpreter could increase the length of time it takes to complete a dietary food recall thus, possibly skewing the data.
* those with self-reported body mass index (BMI) less than the 5th or greater than the 85th percentile (as determined during telephone screen)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy male and female adolescents, ages 12-17 years.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Reporting decay | 6 weeks
  Change (decline) in self-reported energy intake and number of foods consumed over the six-week study duration (Aim 2)
Method preference | 2 weeks
  Participants identify which diet recall method - interviewer-administered or web-based - they prefer overall, and on specific factors, via a qualitative feedback survey at the end of their study involvement (Aim 1)

SECONDARY OUTCOMES:
Feedback on recall methods | 2 or 6 weeks
  Participants in both study aims answer questions about different aspects of using each recall method (Aim 1) or on using their assigned method (Aim 2), such as ease of use, technical challenges, flexibility, duration, and database completeness.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Kalkwarf, PhD, Study Director — Children's Hospital Medical Center, Cincinnati

IPD SHARING:
Plan to Share IPD: No
Not at this time.